CLINICAL TRIAL: NCT06054139
Title: Risk Factors for Refeeding Syndrome in the Surgical Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, serife secgin, Specialist of Anaesthesiology and Reanimation Principle İnvestigator, Samsun University
Other Study IDs: SÜKAEK-2023 12/20
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Refeeding Syndrome
Keywords: hypophosphatemia; hypomagnesemia
MeSH Terms: conditions — Refeeding Syndrome; Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the treated patients in ICU: Patients receiving nutrition while receiving treatment in intensive care
  Interventions: Other: Refeeding Syndrome

INTERVENTIONS:
Other: Refeeding Syndrome — Patients who developed Refeeding Syndrome despite proper nutrition while receiving treatment in the ICU

SUMMARY:
Refeeding Syndrome is a condition that occurs when patients who are undernourished or undernourished suddenly start overfeeding, causing electrolyte disturbances and vitamin deficiencies, resulting in neurological and cardiac problems. It may even result in death. It is aimed to prevent the development of Refeeding Syndrome with nutrition in accordance with the guidelines. The aim of this study is to determine the risk factors for Refeeding Syndrome in Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
Nutritional support is an important part of treatment in intensive care patients. Especially existing comorbidities and developing acute problems before intensive care admission can cause serious malnutrition for patients. Refeeding syndrome is a serious, life-threatening condition accompanied by electrolyte and metabolic disorders as a result of rapid re-feeding following prolonged starvation or malnutrition. The condition may be accompanied by electrolyte disorders such as hypophosphatemia, hypokalemia and hypomagnesemia, as well as decrease in vitamin levels (especially vitamin B1), fluid imbalance and salt retention. The resulting imbalances can cause cardiac and neurological side effects, impaired organ functions and even death. The refeeding protocol should be individualized to each patient's clinical situation. In this study, although nutritional protocols in accordance with the guidelines are applied in patients with risk factors for the development of Refeeding Syndrome, whether Refeeding Syndrome develops and the facilitating factors will be investigated in ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are intensive care patients
2. Patients' age > 18 -

Exclusion Criteria:

1. Diabetic ketoacidosis
2. Other risk factors for hypophosphatemia (patients on continuous hemodialysis, hyperphosphatemia treatment, parathyroidectomy)
3. Patients with pre-study hypophosphatemia (< 0.65 mmol/L)
4. Patients with hyperparathyroidism
5. Terminal stage cancer patients
6. Patients with Glasgow Coma Scale ≤5
7. Patients with respiratory and metabolic alkalosis -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving treatment in intensive care at Samsun University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-07-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Refeeding Syndrome | from june 9, 2023 to june 9, 2024
  Occurrence of RFS：Within 72 hours after feeding serum phosphorus < 0.0.87mmol/L, or from the baseline levels drop > 0.16% or drop > 30%;And (or) hypokalemia, hypomagnesemia, hypocalcemia and corresponding clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGÜR KÖMÜRCÜ, Study Director — SAMSUN UNIVERSITY HOSPITAL
Locations (1):
- Şerife Seçgin, Samsun, Turkey (Türkiye)